CLINICAL TRIAL: NCT05132036
Title: Lung Ultrasound Assessment of Fluid Overload in Haemodialysis Patients Using 8 Sites Score
Brief Title: Lung Ultrasound Assessment of Fluid Overload in Haemodialysis Patients
Acronym: EP8SH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0136
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Lung Ultrasound; Hemodialysis Complication
Keywords: Lung ultrasound; Hemodialysis Complication; hemodialysis ultrafiltration volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lung ultrasound — Subjects are enrolled during their usual session in the hemodialysis unit of the Amiens University Hospital. Before starting the hemodialysis, lung ultrasound according to the "8 sites" score and a measure of bioimpedance will be performed in dorsal decubitus. In a 2nd time, an echocardiography is realized. During haemodialysis session, biological analysis and clinical score will be assessed

SUMMARY:
Determination of the hemodialysis ultrafiltration volume is guided by the clinician's estimate of dry weight. A poor estimate of this dry weight may result in insufficient fluid depletion causing a state of volume overload, which may be associated with long-term left ventricular failure, high blood pressure and excess of mortality. The diagnosis of fluid overload in haemodialysis patient is routinely based on clinical examination which consists of cardiopulmonary auscultation and edema palpation of limb member. Clinical examination can be completed by paraclinical examinations, and bioimpedance is an objective tool that assess fluid overload state. This test provides an individualized hydration status and fluid overload based on normal extracellular volume considering body composition. Echocardiography allows an accurate assessment of blood volume status by simultaneous studying left ventricular filling pressures, systolic pulmonary artery pressure and the diameter of the inferior vena cava. Lung ultrasound analyses the B-lines defined as artefactual images resulting from contact between air in "alveoli" and water in "septa". It can estimate pulmonary congestion. The aim of the study is to evaluate the lung ultrasound using "8 sites" score accuracy for estimating fluid overload of patients before hemodialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* patients on hemodialysis for more than 3 months;
* patients without cardiological or infectious event for at least 3 months;
* patients having at least 2 dialysis session per week;
* patients affiliated with a health insurance plan;
* patients having signed an informed consent.

Exclusion Criteria:

* Pulmonary fibrosis or active lung disease;
* residual diuresis over 500 mL per day;
* body mass index (BMI) < 21 and > 28 Kg/m²;
* medical history of major amputation (subgonal or transfemoral);
* pacemaker carrier;
* patients with orthopedic prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
number of patients with fluid overload | one day
  Fluid overloaded are determined by both tecniques : estimated fluid overload and lung ultrasound measured fluid overload

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No